CLINICAL TRIAL: NCT00285389
Title: Treatment in First Line of Mantle Cell Lymphoma for Patients Under 66 Years by the VAD-CHLORAMBUCIL -Rituximab Regimen Followed by Intensification and Autologous PBSC Transplantation After Marrow Purging With Rituximab
Brief Title: Treatment of Mantle Cell Lymphoma at Diagnosis for Patients Under 65 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Dr Remy GRESSIN Principal Investigator, GOELAMS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MANTEAU 2001
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Chemotherapy; Autologous PBSCT; Molecular evaluation
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Doxorubicin; Dexamethasone; Chlorambucil; Rituximab; Cyclophosphamide; Melphalan; Whole-Body Irradiation; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VAD Clorambucil Rituximab (Experimental)
  Interventions: Drug: Adriblastin; Drug: dexamethasone; Drug: Chlorambucil; Drug: rituximab; Drug: cyclophosphamide; Drug: alkeran; Procedure: Total body irradiation (8Gy/4fr); Drug: vincristine

INTERVENTIONS:
Drug: Adriblastin
Drug: dexamethasone
Drug: Chlorambucil
Drug: rituximab
Drug: cyclophosphamide
Drug: alkeran
Procedure: Total body irradiation (8Gy/4fr)
Drug: vincristine — 0,4 mg/day day 1 to day 4

SUMMARY:
Phase II study to test in first line the VAD (Vincristine Adriablastine Dexamethasone) + C (Chlorambucil ) regimen associated to rituximab ( R-VAD + C ) in a cohort of young patients under 66 years with a mantle cell lymphoma and also the test the role of an in vivo marrow purge with rituximab before an autologous stem cell transplantation for the consolidation of the patients which fulfilled a response to 4 cycles of (R VAD + C) regimen.

DETAILED DESCRIPTION:
All patients at diagnosis with a stage II, III or IV an arbor disease are treated with 4 cycles of (R VAD +C) .

The responders more than RP > 50% received 2 other cycles before to be intensified with alkeran 140 mg/ m2 and a 8 grays TBI over 4 days before an autologous PBSCT.The stem cell collection is realised after a mobilisation with HD Cyclophosphamide (4 mg/m2) after the four R-(VAD + C) cycles and purged by a rituximab injection 10 days before the collection.

There is an clinical and molecular evaluation of the strategy

ELIGIBILITY:
Inclusion Criteria:

* Mantel cell lymphoma
* CD 20+
* At diagnosis or without anterior chemotherapy
* Age >18 and < 66 years
* Ann Arbor ii, III or IV
* ECOG <3
* contraindication for rituximab treatment
* Informed consent signed
* No cancer anteriory
* Renal and hepatic function compatible with the treatment
* Ventricular Fraction > 50 % with echographic method and > 40% with isotopic method

Exclusion Criteria:

* Other type of lymphoma
* age<18 ou > 66 years
* Informed consent not signed
* anterior cancer
* Contraindication to rituximab
* Cardiac insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2002-02; Primary Completion 2005-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
failure event free survival at 3 years | 3 YEARS

SECONDARY OUTCOMES:
Response rate after 4 R-(VAD+C) cycles | 4 months
Incident of Molecular residual disease on blood, marrow and stem cell collection | 3 years
Safety of the R-( VAD+C) regimen | 8 months
Overall survival | 3 years
Efficacy of the stem cell collection after HD Cyclosphosphamide mobilization and rituximab purging | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Remy GRESSIN, MD, Principal Investigator — French Innovative Leukemia Organisation
Locations (3):
- France (3):
  - Regional university hospital, Besançon
  - Regional university hospital, Rennes
  - REgional Hospital, Tours

REFERENCES:
- [Derived] Gressin R, Caulet-Maugendre S, Deconinck E, Tournilhac O, Gyan E, Moles MP, El Yamani A, Cornillon J, Rossi JF, Le Gouill S, Lepeu G, Damaj G, Celigny PS, Maisonneuve H, Corront B, Vilque JP, Casassus P, Lamy T, Colonna M, Colombat P; French GOELAMS Group. Evaluation of the (R)VAD+C regimen for the treatment of newly diagnosed mantle cell lymphoma. Combined results of two prospective phase II trials from the French GOELAMS group. Haematologica. 2010 Aug;95(8):1350-7. doi: 10.3324/haematol.2009.011759. Epub 2010 Mar 10. PMID 20220059